CLINICAL TRIAL: NCT00837642
Title: Vascular Dysfunction in Offspring of Assisted Reproduction Technologies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Urs Scherrer, Professor, University of Lausanne Hospitals
Other Study IDs: 35/07
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Infertility
Keywords: Vascular function in offspring of ART
MeSH Terms: conditions — Infertility | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ART (Assited reproductive technologies): In participants born after IVF will be performed a transthoracic echocardiography
  Interventions: Diagnostic Test: Transthoracic echocardiography
- Control: In participants naturally conceived will be performed a transthoracic echocardiography
  Interventions: Diagnostic Test: Transthoracic echocardiography

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiography — Full transthoracic echocardiography will be performed.

SUMMARY:
The prevalence of infertility has been estimated at 9% worldwide. The steadily increasing use of assisted reproductive technologies (ART) has allowed millions of infertile couples to have children. These children make up for 1 to 4% of the population in developed countries. ART involves the manipulation of early embryos at a time when they may be particularly vulnerable to external disturbances. In line with this concept, studies in mice suggest that ART alters the activity of enzymes involved in the regulation of metabolic and cardiovascular homeostasis. Alternatively, infertility itself or the drugs used to stimulate ovulation may have adverse effects on the outcome of the offspring. The safety of ART for long-term health is, therefore, of utmost importance. Among the potential long-term consequences of ART, cardiovascular disease may represent an important candidate, but there is no information.

Investigators show that, children born after in vitro fertilization (IVF) present systemic and pulmonary vascular dysfunction at high-altitude when compared to age- and sex-matched control subjects. A 5 years follow-up study shows that premature vascular aegieng persist and evolve to arterial hypertension. Arterial hypertension may induce cardiac dysfunction.

Therefore, the major goal of this proposal is to assess cardiac function in apparently healthy participants born after ART.

ELIGIBILITY:
Inclusion Criteria:

* Offspring of ART
* Healthy
* Born at term

Exclusion Criteria:

* Cardio-pulmonary malformations
* Neuro-muscular malformations

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All the partcicipants that have been participated in our previous studies will be asked to take part in this new study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-10; Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Cardiac function | 1 year
  Ejection fraction [%]

SECONDARY OUTCOMES:
Left ventricular musce mass | 1 year
  Left ventricular muscle mass [g/m2]

CONTACTS AND LOCATIONS:
Overall Officials: Emrush Rexhaj, PD, Principal Investigator — University Hospital of Bern, Cardiology, Switzerland
Locations (1):
- University Hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] Meister TA, Rimoldi SF, Soria R, von Arx R, Messerli FH, Sartori C, Scherrer U, Rexhaj E. Association of Assisted Reproductive Technologies With Arterial Hypertension During Adolescence. J Am Coll Cardiol. 2018 Sep 11;72(11):1267-1274. doi: 10.1016/j.jacc.2018.06.060. PMID 30190005
- [Derived] Scherrer U, Rimoldi SF, Rexhaj E, Stuber T, Duplain H, Garcin S, de Marchi SF, Nicod P, Germond M, Allemann Y, Sartori C. Systemic and pulmonary vascular dysfunction in children conceived by assisted reproductive technologies. Circulation. 2012 Apr 17;125(15):1890-6. doi: 10.1161/CIRCULATIONAHA.111.071183. Epub 2012 Mar 20. PMID 22434595